CLINICAL TRIAL: NCT05183399
Title: Treatment of Patients With Traumatic or Iatrogenic Vessel Injuries in Thoracic, Abdominal, and Pelvic Arteries
Brief Title: Treatment of Patients With Traumatic or Iatrogenic Vessel Injuries
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: JPS 16-04
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Iatrogenic Vessel Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: GORE® VIABAHN® Endoprosthesis

SUMMARY:
The purpose of this study is to confirm device efficacy and safety of the GORE® VIABAHN® Endoprosthesis (hereafter "VB device") for the treatment of traumatic or iatrogenic vessel injury in thoracic, abdominal, and pelvic arteries (except the aorta, coronary, brachiocephalic, carotid, vertebral and pulmonary arteries).

ELIGIBILITY:
Patients with traumatic or iatrogenic vessel injuries in thoracic, abdominal, and pelvic arteries (except the aorta, coronary, brachiocephalic, carotid, vertebral and pulmonary arteries ) with a reference vessel diameter ranging from 4.0 to 12.0mm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with traumatic or iatrogenic vessel injuries in thoracic, abdominal, and pelvic arteries (except the aorta, coronary, brachiocephalic, carotid, vertebral and pulmonary arteries ) with a reference vessel diameter ranging from 4.0 to 12.0mm.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
Technical Success | Day 1 to 1 Month
  A technical success is defined as is a successful device implantation and a successful hemostasis.

SECONDARY OUTCOMES:
Safety | Day 1 to 12 months
  The safety Endpoint is the occurrence of serious adverse events and deficiencies.